CLINICAL TRIAL: NCT05897541
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of S-217622 in the Prevention of Symptomatic SARS-CoV-2 Infection in Household Contacts of an Individual With Symptomatic COVID-19
Brief Title: Phase 3 Study of S-217622 in Prevention of Symptomatic SARS-CoV-2 Infection
Acronym: SCORPIO-PEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2206T1331; 2022-002898-28 (EudraCT Number); 2023-503200-91-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2023-06-06; First posted 2023-06-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — ensitrelvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S-217622 (Experimental): S-217622 will be administered orally for 5 days.
  Interventions: Drug: S-217622
- Placebo (Placebo Comparator): Placebo matching to S-217622 will be administered orally for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-217622 — Administered as a tablet.
  Arms: S-217622
Drug: Placebo — Administered as a tablet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the proportion of participants who are infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (positive reverse transcription polymerase chain reaction [RT-PCR] test) and have coronavirus disease 2019 (COVID-19) symptom(s) with S-217622 tablets compared with placebo tablets in participants who are household contacts of an individual with symptomatic COVID-19.

DETAILED DESCRIPTION:
This study will enroll 2 types of participants: 1. those with a negative screening SARS-CoV-2 infection (referred to as "study participants"); 2. those with a positive screening SARS-CoV-2-infection (referred to as "index participants"). Study participants will receive study intervention (S-217622 or placebo), index participants will receive no study intervention.

ELIGIBILITY:
Inclusion Criteria:

Index Participants

Only 1 index participant from each household will be enrolled in the study. Participants are eligible to be included as an index participant if all of the following criteria apply:

1. Pediatric participants or adult participants (of any age)
2. The index participant must:

   1. Have at least 1 COVID-19 symptom within 24 hours before the index participant providing informed consent. COVID-19 symptom(s) must be deemed by the investigator as related to the current SARS-CoV-2 infection (not related to preexisting comorbidities) or deemed as preexisting and worsened due to SARS-CoV-2 infection.
   2. Must have positive SARS-CoV-2 test (a nucleic acid amplification test or antigen test) from any respiratory tract specimen from a sample collected prior to randomization of the participant
3. Must have a potential study participant who can participate in the study after onset of COVID-19 symptoms in an index participant

Study Participants

Multiple study participants from the same household are allowed to be enrolled in the study. The study intervention randomization will be performed based at the study participant's level. Participants will be eligible to be included in the study only if all of the following criteria apply:

1. ≥ 12 years of age at the time of signing the informed consent
2. Has a negative screening for SARS-CoV-2 infection, as determined by SARS-CoV-2 test (a nucleic acid amplification test or antigen test) from any respiratory tract specimen (for example, oropharyngeal, nasopharyngeal or nasal swab, or saliva).
3. Has lived in household with index participant and will continue to live in same household and share common areas such as dining rooms and bathrooms until the end of the study
4. Must not be considered by the investigator or subinvestigator to have SARS-CoV-2 infection and:

   1. No measured fever at Screening (defined as body temperature ≥ 38.0°Celsius [C] per tympanic or rectal thermometer or ≥ 37.5°C per axillary, oral, or forehead/temporal thermometer)
   2. No COVID-19 symptoms at Screening (if a participant has COVID-19-like symptoms caused by comorbidities, only 1 symptom will be allowed)
5. Capable and willing to complete a participant diary
6. a. Male participants: Participants with partners that are woman of childbearing potential (WOCBP) must agree to use effective contraception. Participants with pregnant partners must agree to use effective contraception.

   b. Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and the following conditions applies:
   * Is not a WOCBP or
   * All of the following apply:

     * Is a WOCBP and using a contraceptive method that is effective as described in the protocol.
     * A WOCBP must have a negative urine pregnancy test within 24 hours before the first dose of study intervention period.
     * If a urine pregnancy test cannot be confirmed as negative (for example, an ambiguous result), a serum pregnancy test must be negative.
   * Additional requirements for pregnancy testing during and after study intervention as described in the protocol.
   * The investigator/subinvestigator will review medical history, menstrual history, and recent sexual activity to decrease the risk of inclusion of a woman with an early undetected pregnancy.
7. Participant must be randomized ≤ 72 hours from onset of COVID-19 symptoms in the index participant.

Exclusion Criteria:

Study Participants: Participants will be excluded from the study if any of the following criteria apply:

1. Tested positive for SARS-CoV-2 in the past 6 months.
2. Have an underlying disease requiring systemic corticosteroids (excluding topical), antipyretics/analgesics, or immunosuppressive agents.
3. Known current renal impairment defined as creatinine clearance < 30 milliliters/minute by Cockcroft Gault or requiring dialysis.
4. Participants with severe liver dysfunction, such as known history of cirrhosis or liver decompensation (including ascites, variceal bleeding, or hepatic encephalopathy).
5. Received approved, authorized, or investigational convalescent plasma, or other anti- SARS-CoV-2 biologic products within 3 months of the Screening Visit
6. Received approved, authorized, or investigational anti-SARS-CoV-2 monoclonal antibodies (mAbs) in the last 6 months.
7. Received any SARS-CoV-2 vaccine within 6 months prior to the Screening Visit or is expected to receive a SARS-CoV-2 vaccine or other approved, authorized, or investigational postexposure prophylaxis treatments until the end of the study.
8. Participants who have used any of the following drugs within 14 days prior to enrollment:

   1. Strong cytochrome P450 (CYP) 3A inducer
   2. Products containing St. John's wort
9. Exposed to an investigational drug within 30 days or 5 half-lives of the drug prior to the Screening Visit.
10. Positive urine pregnancy test at Screening Visit or are lactating.
11. Known allergy/sensitivity or any hypersensitivity to components of S-217622 or placebo for S-217622.
12. Any condition or circumstance that, in the opinion of the investigator or subinvestigator, would compromise the safety of the participant or the quality of the study data.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2387 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants in the Modified Intention-to-treat (mITT) Population with a Negative Screening SARS-CoV-2 Infection who are Infected with SARS-CoV-2 and Have COVID-19 Symptoms Onset | Day 1 through Day 10

SECONDARY OUTCOMES:
Number of Participants in the Intention-to-treat (ITT) Population with a Negative Screening SARS-CoV-2 Infection who are Infected with SARS-CoV-2 and Have COVID-19 Symptoms Onset | Day 1 through Day 10
Number of Participants Infected with SARS-CoV-2 Regardless of Occurrence of COVID-19 Symptoms | Day 1 through Days 10, 15, or 28
Time to the First Positive RT-PCR Result | Day 1 through Day 10
Number of Participants with a Positive RT-PCR Result | Day 1 through Day 10
Number of Participants Infected with SARS-CoV-2 with no COVID-19 Symptoms | Day 1 through Day 10
Number of Participants with Sustained Resolution of all COVID-19 Symptoms | Day 1 through Day 28
Number of Participants with Sustained Resolution of Each COVID-19 Symptom | Day 1 through Day 28
Change in Total Score of COVID-19 Symptoms | Day 1 through Day 10
Time From First Confirmed SARS-CoV-2 Until at Least 1 COVID-19 Symptom | Day 1 through Day 28
Time From First Confirmed SARS-CoV-2 Until COVID-19 Symptoms Onset | Day 1 through Day 28
Number of Participants Experiencing Hospitalization or Death from Any Cause | Day 1 through Day 28
Plasma Concentration of S-217622 | Day 3, Day 6, and Event Driven
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 28

CONTACTS AND LOCATIONS:
Locations (178):
- United States (95):
  - Central Alabama Research, Birmingham, Alabama
  - Accel Research Site - Achieve - Birmingham - ERN - PPDS, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Absolute Clinical Research, LLC, Phoenix, Arizona
  - One of a Kind Clinical Research Center LLC, Scottsdale, Arizona
  - Healthstar Research, Hot Springs, Arkansas
  - Preferred Research Partners - ClinEdge - PPDS, Little Rock, Arkansas
  - Neighborhood Healthcare, Escondido, California
  - Apex Research Group, Fair Oaks, California
  - Ascada Research LLC, Fullerton, California
  - Torrance Clinical Research Institute, Lomita, California
  - Ark Clinical Research - Long Beach - ClinEdge - PPDS, Long Beach, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Smart Cures Clinical Research, Rolling Hills Estates, California
  - Clinical Trials Management Services, LLC, Thousand Oaks, California
  - Lynn Institute of The Rockies - ERN - PPDS, Colorado Springs, Colorado
  - TrueBlue Clinical Research, Brandon, Florida
  - Invictus Clinical Research Group, LLC, Coconut Creek, Florida
  - Universal Medical and Research Center, LLC, Coral Gables, Florida
  - Hope Clinical Trials, Coral Gables, Florida
  - I.V.A.M. Clinical & Investigational Center, Doral, Florida
  - Quality Research of South Florida, Hialeah, Florida
  - Universal Medical and Research Center, LLC Homestead, Homestead, Florida
  - Flourish Research - Leesburg - PPDS, Leesburg, Florida
  - Premier Clinical Research Institute - Miami - ClinEdge - PPDS, Miami, Florida
  - LCC Medical Research - Miami - ClinEdge - PPDS, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Suncoast Research Group LLC - Flourish - PPDS, Miami, Florida
  - University of Miami - 1150 NW 14th St, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Oceane7 Medical & Research Center, Inc., Miami, Florida
  - Continental Clinical Research, LLC, Miami, Florida
  - BioClinical Research Alliance, Miami, Florida
  - Ivetmar Medical Group, LLC, Miami, Florida
  - Miami Clinical Research - ClinEdge - PPDS, Miami, Florida
  - Global Health Clinical Trials, Miami, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Alma Research, Miami, Florida
  - GCP Global Clinical Professionals, LLC, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Kendall South Medical Center, Miami, Florida
  - Flourish Research - Miami - PPDS, Miami, Florida
  - Meridian International Research, Miami Lakes, Florida
  - MedQuest Translational Sciences, Miami Lakes, Florida
  - Combined Research Orlando Phase I-IV LLC, Orlando, Florida
  - Central Florida Internists - Conway, Orlando, Florida
  - Accel Research Sites - Nona Pediatric Center - ERN - PPDS, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - CTMD Research, Inc. Palm Springs - Hunt - PPDS, Palm Springs, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Progressive Medical Research - ClinEdge - PPDS, Port Orange, Florida
  - Renew Health Clinical Research, LLC, Tampa, Florida
  - Bayside Clinical Research-West Tampa, Tampa, Florida
  - Tampa Bay Health Care, Tampa, Florida
  - Balanced Life Health Care Solutions - SKYCRNG - PPDS, Lawrenceville, Georgia
  - Olivo Medical and Wellness Center, Chicago, Illinois
  - Eagle Clinical Research, Chicago, Illinois
  - KU Wichita Center for Clinical Research, Wichita, Kansas
  - Voyage Medical - Michigan, Canton, Michigan
  - Vida Clinical Sites, Dearborn Heights, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Velocity Clinical Research - Covington - PPDS, Gulfport, Mississippi
  - Montana Medical Research, Missoula, Montana
  - Child Healthcare Associates - East Syracuse, East Syracuse, New York
  - Rochester Clinical Research - ATLAS - Rochester - PPDS, Rochester, New York
  - Lapis Clinical Research-Denver, Denver, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - WellNow Urgent Care & Research - Huber Heights, Dayton, Ohio
  - PriMed Clinical Research - ClinEdge - PPDS, Dayton, Ohio
  - Cyn3rgy Research - ClinEdge - PPDS, Gresham, Oregon
  - Tristar Clinical Investigations, P.C., Philadelphia, Pennsylvania
  - Frontier Clinical Research - Scottdale, Scottdale, Pennsylvania
  - Coastal Pediatric Associates, Charleston, South Carolina
  - SPICA Clinical Research, Columbia, South Carolina
  - Main Street Physicians Care - Waterway, Little River, South Carolina
  - Clinical Trials of South Carolina - ClinEdge - PPDS, Moncks Corner, South Carolina
  - Saint Hope Foundation Inc, Bellaire, Texas
  - ACRC Trials - Carrollton - Hunt - PPDS, Carrollton, Texas
  - Global Medical Research - M3 WR, Dallas, Texas
  - Alina Clinical Trials, LLC, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Epic Medical Research LLC - DeSoto, DeSoto, Texas
  - Care United Research, LLC - Elligo - PPDS, Forney, Texas
  - Valley Institute of Research, Fort Worth, Texas
  - C & R Research Services USA, Houston, Texas
  - New Horizon Medical Group, LLC, Houston, Texas
  - Care and Cure Clinic, Houston, Texas
  - DCT-McAllen Primary Care Research, LLC dba Discove, McAllen, Texas
  - Advances In Health Inc, Pearland, Texas
  - Clinical Associates in Research Therapeutics of America, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Alliance for Multispecialty Research, LLC - Kaysville - PPDS, Kaysville, Utah
  - Alliance for Multispecialty Research LLC - Roy, Roy, Utah
- Argentina (11):
  - Hospital Interzonal General de Agudos Vicente Lopez Y Planes, General Rodríguez, Buenos Aires
  - Clínica Privada Independencia, Munro, Buenos Aires
  - Centro Médico San Nicolás Grupo Oroño, San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clínicas Zárate, Zárate, Buenos Aires
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario, Santa Fe Province
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - Hospital Rawson, Córdoba
  - Sanatorio Allende S.A, Córdoba
  - Sanatorio Medico de Diagnostico Y Tratamiento, Santa Fe
- Japan (67):
  - Kamezawa Clinic, Kasugai-Shi, Aiti
  - Hosokawa Surgical Clinic, Nagoya-Shi Nakamura-Ku, Aiti
  - Fujimaki Ear, Nose and Throat Clinic (Ent Clinic), Ichikawa-Shi, Chiba
  - Tomita Internal medicine clinic, Fukuoka, Fukuoka
  - Irie Naika Syounika Iin, Fukuoka, Fukuoka
  - Tashiro Endocrinolgy Clinic, Fukuoka, Fukuoka
  - Megumi Clinic, Kasuyagun Shimemachi, Fukuoka
  - Suto Hospital, Annaka-shi, Gunma
  - Shoda Hospital, Annaka-Shi, Gunma
  - Uno Internal Medicine Respiratory Clinic, Isesaki-Shi, Gunma
  - Kikuchi Internal clinic, Maebashi, Gunma
  - Teine Otolaryngology Clinic, Sapporo, Hokkaidô
  - Maruyama Tame Pediatrics, Sapporo, Hokkaidô
  - Nishioka Hospital, Sapporo-Shi Toyohira-Ku, Hokkaidô
  - Japanese Red Cross Fukuoka Hospital, Fukuoka, Hukuoka Province
  - Iizuka Hospital, Iizuka-Shi, Hukuoka
  - Morizono medical clinic, Kitakyushu-shi, Hukuoka
  - Nagata Hospital, Yanagawa-Shi, Hukuoka
  - Toda Internal Medicine ＆ Neurology, Akashi-Shi, Hyôgo
  - Terada Clinic Respiratory Medicine and General Practice, Himeji-shi, Hyôgo
  - Takahashi Pediatric Clinic, Kobe-Shi Nada-Ku, Hyôgo
  - Nishiyamato Keiwa Hospital, Naka, Ibaraki
  - Hitachi,Ltd.,Tsuchiura Medical & Health Care Center, Tsuchiura, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura-Shi, Ibaraki
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Moriyama Otolaryngology, Kagoshima, Kagoshima-ken
  - Kamoike Otolaryngology Clinic, Kagoshima, Kagoshima-ken
  - Murasakibaru Tahara Hospital, Kagoshima, Kagoshima-ken
  - Motosumiyoshi-ekimae Cocoromi Clinic, Kawasaki-Shi, Kanagawa
  - Kanagawa Himawari Clinic, Kawasaki-Shi, Kanagawa
  - Medical Corporation Nakano Children's Clinic, Yokohama, Kanagawa
  - Kaiseikai Kita Shin Yokohama Internal Medicine Clinic, Yokohama, Kanagawa
  - Yokohama Municipal Citizens Hospital, Yokohama, Kanagawa
  - Nagaoka Chuo General Hospital, Nagaoka-Shi, Niigata
  - NHO Okinawa Hospital, Ginowan-Shi, Okinawa
  - University of the Ryukyus Hospital - 207 Uehara, Okinawa-Shi, Okinawa
  - Rinku General Medical Center, Izumisano, Osaka
  - Lee's Clinic, Osaka, Osaka
  - Kasukabe Medical Center, Kasukabe, Saitama
  - Fujimino Emergency Hospital, Miyoshi-machi, Iruma-gun, Saitama
  - Fukuda Medical Clinic, Toda-shi, Saitama
  - KODAIRA Hospital, Toda-Shi, Saitama
  - Medical Corporation Kojyokai Hirose Clinic, Tokorozawa-Shi, Saitama
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - Global Healthcare Clinic, Chiyoda-Ku, Tokyo
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - Nishikasai ekimae Family Clinic, Edogawa-ku, Tokyo
  - Takinogawa Hospital, Kita-ku, Tokyo
  - Musashino Hospital, Kodaira-Shi, Tokyo
  - Takahashi Medical Clinic, Kokubunji-Shi, Tokyo
  - Nozaki Clinical, Musashino-Shi, Tokyo
  - Shimamura Memorial Hospital, Nerima-Ku, Tokyo
  - MIH Clinic Yoyogi, Shibuya-Ku, Tokyo
  - Tokyo Shinagawa Hospital Social Medical Corporation Association Tokyokyojuno-kai, Shinagawa-ku, Tokyo
  - Yotsuya Naika, Shinjuku-Ku, Tokyo
  - Yoshida Clinic, Suginami-ku, Tokyo
  - Denenchofu Family Clinic, Ōta-ku, Tokyo Province
  - Toyama Rosai Hospital, Uozu-Shi, Toyama
  - Kijima Kids Clinic, Higashiokitama-gun, Yamagata
  - Nakayama Pediatric Clinic, Nagasaki
  - Okayama University Hospital, Okayama
  - Osaka City Juso Hospital, Osaka
  - Soyukai Medical Corporation Yamaguchi clinic, Ōta-ku
  - Shiwa Chuo Syounika, Shiwa-gun
  - Shizuka Medical Clinic, Takasaki-shi
  - Ikebukuro Higashiguchi Mame Clinic, Toshima-ku
  - Suita Municipal Hospital, Suita, Ôsaka
- South Africa (3):
  - Newtown Clinical Research Centre, City of Johannesburg, Gauteng
  - NMMM PHARMEDICA Health Research Institute, Lombardy East, Johannesburg, Gauteng
  - Trident Clinical, Sol Plaatjie, Northern Cape
- Vietnam (2):
  - Hanoi University of Medicine - Clinical Trial Unit, Quận Đống Đa, Ha Noi, Thu Do
  - University of Medicine Center, Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No